CLINICAL TRIAL: NCT04698512
Title: MAgic Touch™ Intervention Leap for Dialysis Access (MATILDA) Trial
Brief Title: MAgicTouch™ Intervention Leap for Dialysis Access (MATILDA) Trial
Acronym: MATILDA
Status: Completed | Type: Observational
Sponsor: Singapore General Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: MATILDA
Record Dates: First submitted 2020-12-28; First posted 2021-01-07 (Actual); Last update posted 2021-03-17 (Actual); Status verified 2021-03

CONDITIONS: Dialysis Access Malfunction; End Stage Renal Failure on Dialysis; End Stage Renal Disease; Fistulas Arteriovenous; Stenosis
Keywords: Sirolimus coated balloon; Target lesion primary patency; Arterio-venous fistula; Outcome; Safety
MeSH Terms: conditions — Kidney Failure, Chronic; Arteriovenous Fistula; Constriction, Pathologic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Arteriovenous Fistuloplasty with MagicTouch™ Balloon: Patients above the age of 21 that have undergone AVF / AVG fistuloplasty with MagicTouch™ at Singapore General Hospital will be included in the study and followed up post-op for 12 months. Patients will be treated and followed-up following standard clinical care pathways.
  Interventions: Device: AVFistuloplasty with Sirolimus coated balloon

INTERVENTIONS:
Device: AVFistuloplasty with Sirolimus coated balloon — After an initial fistulogram, the lesion will first be predicated with standard high pressure balloon, followed by MagicTouch™ Sirolimus drug coated balloon

SUMMARY:
For patients with End Stage Renal Failure (ESRF), the surgical creation of an Autogenous Arteriovenous Fistula (AVF) or Autogenous Arteriovenous Graft (AVG) is the recognised standard for providing vascular access. A functioning dialysis vascular access is essential to facilitate hemodialysis (HD) treatment. Advantages include improved hemodialysis initiation time, improved dialysis quality, better maintenance of accesses and generally, better outcomes in patients. Unfortunately almost 50% of AVF and AVG fail after a median lifetime of 3 to 7 years and 12 to 18 months respectively. Vascular access dysfunction is a major cause of morbidity and hospitalisation for ESRF patients, costing the healthcare system USD 18 million globally. Venous stenosis and scarring are caused by trauma from surgical access creation when the circuit comes arterialized and from repeated percutaneous punctures from subsequent hemodialysis. This study is performed to evaluate Sirolimus-coated balloon efficacy and safety using MagicTouch™ Drug coated balloon catheter (Concept Medical Inc, Tampa, FL, US) on AVF patency with de novo and recurrent stenosis.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent was obtained
* Patient aged ≥ 21 and ≤ 90 years
* Native AVF was created more than 2 months prior to index procedure and had undergone 10 or more haemodialysis sessions utilizing two needles
* Target lesion location had to be located between the anastomoses to the axillary-subclavian vein junction, as defined by insertion of the cephalic vein
* On initial fistulogram, target lesions stenosis had to be ≥50 on angiographic assessment and in keeping with the clinical indicator for intervention
* Stenosis had to <12cm in length (to allow for potential treatment with one SCB (length 15cm) only
* Stenosis had to be initially treated successfully with a high-pressure plain balloon prior to SCB treatment as defined by:- (A) no clinically significant dissection (flow limiting) (B) no extravasation requiring treatment/stenting (C) residual stenosis ≤30% by angiographic measurement (D) Ability to completely efface the lesion waist using the pre-dilation balloon
* No more than one additional ("nontarget") lesion in the access circuit that had to be also successfully treated (≤30% residual stenosis) before drug elution. Separate lesion was defined by at least 3cm in distance from the target lesion.
* Reference vessel diameter 5mm-8mm

Exclusion Criteria:

* Women who were preganant, lactating, or planning on becoming pregnant during the study
* Subject had more than 2 lesions in the access circuit
* Subject had a secondary non-target lesion that could not be successfully treated
* Sepsis or active infection
* Asymptomatic target lesions
* A thrombosed access or an access with thrombosis treated ≤ 30 days prior to index procedure
* Surgical revision of the access site performed, planned or expected ≤ 3months before or after the index procedure
* Patients who were taking immunosuppressive therapy or are routinely taking ≥15 mg prednisone per day
* Currently participating in another investigational drug, biologic, or device study involving Sirolimus or paclitaxel
* Contraindication to Aspirin or Clopidogrel usage
* Mental condition rendering the subject unable to understand the nature, scope and possible consequences of the study, or language barrier such that the subject is unable to give informed consent
* Uncooperative attitude or potential for non-compliance with the requirements of the protocol making study participation impractical
* Where final angioplasty treatment requires a stent or drug eluting balloon >8mm in diameter
* Metastatic cancer or terminal medical condition
* Blood coagulation disorders
* Limited life expectancy (<12 months)
* Allergy or other know contraindication to iodinated media contrast, heparin, or Sirolimus

Ages: 21 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who have received inpatient treatment (i.e. fistuloplasty) for their failing dialysis access at Singapore General Hospital
Sampling Method: Non-Probability Sample
Enrollment: 35 (Actual)
Dates: Start 2019-05-21 (Actual); Primary Completion 2020-01-16 (Actual); Study Completion 2021-01-30 (Actual)

PRIMARY OUTCOMES:
Target Lesion Primary Patency | 3-months post op
  No need for clinically driven reintervention of target lesion, no access thrombosis and no significant restenosis (lumen diameter <2.7mm) on duplex ultrasound
Target Lesion Primary Patency | 6-months post op
  No need for clinically driven reintervention of target lesion, no access thrombosis and no significant restenosis (lumen diameter <2.7mm) on duplex ultrasound
Freedom from localised or systemic serious adverse events | 30 days post-op
  Include life-threatening events or those resulting in death, requiring hospitalisation, resulting in permanent disability, or requiring intervention to prevent permanent impairment

SECONDARY OUTCOMES:
Access circuit patency | 3 and 6 months post op
  Lack of stenosis in any region of the AVF circuit requiring intervention
Procedural success | Day of operation
  Defined as technical success with at least one indicator of hemodynamic or clinical success. I.e. no conduit rupture during any of the procedures requiring bailout stenting.
Primary assisted patency | 3 and 6 months post op
  Lack of access circuit thrombosis requiring thrombolysis
Number of open bypass revision surgery required to maintain access circuit primary patency | 3 and 6 months post op
Secondary access patency | 3 and 6 months post-op
  Lack of dialysis access abandonment
Number of interventions required to maintain access circuit primary patency | 3 and 6 months post-op
Event of mortality | 6 months post-op

CONTACTS AND LOCATIONS:
Overall Officials: Tjun Yip Tang, Principal Investigator — Singapore General Hospital
Locations (1):
- Singapore General Hospital, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lee T, Roy-Chaudhury P. Advances and new frontiers in the pathophysiology of venous neointimal hyperplasia and dialysis access stenosis. Adv Chronic Kidney Dis. 2009 Sep;16(5):329-38. doi: 10.1053/j.ackd.2009.06.009. PMID 19695501
- [Background] Pantelias K, Grapsa E. Vascular access today. World J Nephrol. 2012 Jun 6;1(3):69-78. doi: 10.5527/wjn.v1.i3.69. PMID 24175244